CLINICAL TRIAL: NCT04606732
Title: Cardiovascular Clinical Features and Cardiovascular Therapies in the Development, Progression and Outcome of Patients with SARS-Cov-2 Related Pneumonia
Brief Title: CardioVascular Disease Progression and Prognosis in COVID-19
Acronym: CVP-Covid19
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Olivia Manfrini, MD, MD, University of Bologna
Other Study IDs: CV_SPP_COVID19
Record Dates: First submitted 2020-10-27; First posted 2020-10-28 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Covid19
Keywords: Cardiovascular Diseases; Pneumonia, Viral; SARS-CoV-2; Covid-12; ACE receptor
MeSH Terms: conditions — COVID-19; Cardiovascular Diseases; Pneumonia, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The CVP-COVID19 registry is both a retrospective and prospective study design in order to identify predictors of cardiovascular disease progression and mortality for COVID-19. The registry enrolls consecutive patients with positive microbiological tests for SARS-CoV-2 admitted to an academic hospital in northern Italy for worsening of COVID-19 symptoms. The study does not test any new diagnostic or therapeutic approach. Patients are treated according to good clinical practice. Patients characteristics, including medical history (with particular attention to cardiovascular and pneumological risk factors), features of physical examination, results laboratory and radiological tests and treatments (pre- and in-hospital) are related with patient outcome. Logistic analysis (univariate, multivariate and propensity) are performed in order to identify factors associated with disease progression. Primary endpoint: mortality.

DETAILED DESCRIPTION:
Members of the Steering Committee:

Olivia Manfrini (Università di Bologna, Italy) Raffaele Bugiardini (Università di Bologna, Italy) Stefano Nava (Università di Bologna, Italy) Elisabetta Poluzzi (Università di Bologna, Italy) Maria Carla Re (Università di Bologna, Italy) Caterina Vocale (Policlinico Sant'Orsola) Study Coordinator: Edina Cenko (Università di Bologna, Italy)

ELIGIBILITY:
Inclusion Criteria:

hospitalization for COVID-19

Exclusion Criteria:

age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted to an academic hospital in northern Italy for worsening of COVID-19 symptoms
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  All causes mortality
Mortality | 6 months
  All causes mortality
Mortality | 1 year
  All causes mortality

CONTACTS AND LOCATIONS:
Overall Officials: Olivia Manfrini, MD, Principal Investigator — DIMEC, Università di Bologna
Locations (1):
- Policlinico Sant'Orsola, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bergami M, Manfrini O, Nava S, Caramori G, Yoon J, Badimon L, Cenko E, David A, Demiri I, Dorobantu M, Fabin N, Gheorghe-Fronea O, Jankovic R, Kedev S, Ladjevic N, Lasica R, Loncar G, Mancuso G, Mendieta G, Milicic D, Mjehovic P, Pasalic M, Petrovic M, Poposka L, Scarpone M, Stefanovic M, van der Schaar M, Vasiljevic Z, Vavlukis M, Vega Pittao ML, Vukomanovic V, Zdravkovic M, Bugiardini R. Relationship Between Azithromycin and Cardiovascular Outcomes in Unvaccinated Patients With COVID-19 and Preexisting Cardiovascular Disease. J Am Heart Assoc. 2023 Jul 18;12(14):e028939. doi: 10.1161/JAHA.122.028939. Epub 2023 Jul 14. PMID 37449568
- [Background] Bugiardini R, Nava S, Caramori G, Yoon J, Badimon L, Bergami M, Cenko E, David A, Demiri I, Dorobantu M, Fronea O, Jankovic R, Kedev S, Ladjevic N, Lasica R, Loncar G, Mancuso G, Mendieta G, Milicic D, Mjehovic P, Pasalic M, Petrovic M, Poposka L, Scarpone M, Stefanovic M, van der Schaar M, Vasiljevic Z, Vavlukis M, Vega Pittao ML, Vukomanovic V, Zdravkovic M, Manfrini O. Sex differences and disparities in cardiovascular outcomes of COVID-19. Cardiovasc Res. 2023 May 22;119(5):1190-1201. doi: 10.1093/cvr/cvad011. PMID 36651866
- [Background] Cenko E, Badimon L, Bugiardini R, Claeys MJ, De Luca G, de Wit C, Derumeaux G, Dorobantu M, Duncker DJ, Eringa EC, Gorog DA, Hassager C, Heinzel FR, Huber K, Manfrini O, Milicic D, Oikonomou E, Padro T, Trifunovic-Zamaklar D, Vasiljevic-Pokrajcic Z, Vavlukis M, Vilahur G, Tousoulis D. Cardiovascular disease and COVID-19: a consensus paper from the ESC Working Group on Coronary Pathophysiology & Microcirculation, ESC Working Group on Thrombosis and the Association for Acute CardioVascular Care (ACVC), in collaboration with the European Heart Rhythm Association (EHRA). Cardiovasc Res. 2021 Dec 17;117(14):2705-2729. doi: 10.1093/cvr/cvab298. PMID 34528075